CLINICAL TRIAL: NCT04961918
Title: The Efficacy of Hepatic Arterial Infusion Chemotherapy (HAIC) Combine Lenvatinib and Durvalumab (HILL) in Advanced Hepatocellular Carcinoma (HCC): A Prospective, Single-armed, Stage II Clinical Trial
Brief Title: The Efficacy of Hepatic Arterial Infusion Chemotherapy (HAIC) Combine Lenvatinib and Durvalumab (HILL) in Advanced Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rong-ping Guo, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HILL-001
Record Dates: First submitted 2021-07-13; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Hepatic Arterial Infusion Chemotherapy (HAIC) Combine Lenvatinib and Durvalumab (HILL)
  Interventions: Procedure: Hepatic Arterial Infusion Chemotherapy (HAIC) Combine Lenvatinib and Durvalumab (HILL)

INTERVENTIONS:
Procedure: Hepatic Arterial Infusion Chemotherapy (HAIC) Combine Lenvatinib and Durvalumab (HILL) — Hepatic Arterial Infusion Chemotherapy (HAIC) Combine Lenvatinib and Durvalumab (HILL)

SUMMARY:
To evaluate the efficacy of HAIC combine Lenvatinib and Durvalumab (HILL) in advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old and younger than 75 years; ECOG PS≤1; proven advanced hepatocellular carcinoma according patological examination or EASL/AASLD diagnostic criteria; not previous treated for tumor; cannot accepted hepatectomy; the lab test could meet: neutrophil count≥2.0×109/L; hemoglobin≥100g/L; platelet count≥75×109/L; serum albumin≥35g/L; total bilirubin<2-times upper limit of normal; ALT<3-times upper limit of normal; AST<3-times upper limit of normal; serum creatine<1.5-times upper limit of normal; PT≤upper limit of normal plus 4 seconds; INR≤2.2; sign up consent;

Exclusion Criteria:

* cannot tolerate HAIC or lenvatinib or durvalumab; known history of other malignancy; be allergic to related drugs; underwent organ transplantation before; be treated before (interferon included); known history of HIV infection; known history of drug or alcohol abuse; have GI hemorrhage or cardiac/brain vascular events within 30 days; pregnancy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-07-13 (Estimated); Primary Completion 2022-07-13 (Estimated); Study Completion 2023-07-13 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of progression, assessed up to 36 months
  progression-free survival

SECONDARY OUTCOMES:
ORR | From date of randomization until the date of death, assessed up to 36 months
  objective response rate
DCR | From date of randomization until the date of death, assessed up to 36 months
  disease control rate
OS | From date of randomization until the date of death from any cause, assessed up to 36 months
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- SUN YAT-SEN University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided